CLINICAL TRIAL: NCT03389659
Title: A Randomized, Multicenter, Double-blinded, Phase III Study of Vitamin D3 in Combination With Oxaliplatin Plus Fluoropyrimidine Versus Oxaliplatin Plus Fluoropyrimidine as First-line Chemotherapy in Previously Untreated Advanced or Metastatic Colorectal Cancer
Brief Title: XELOX/mFOLFOX Plus Vitamin D3 vs. XELOX/mFOLFOX as Firstline Chemotherapy in mCRC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TianjinCIH20171212
Record Dates: First submitted 2017-12-14; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Vitamin D3
Keywords: mCRC; oxaliplatin plus fluoropyrimidine
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blined
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 group (Experimental): vitamin D3 2000IU (400IU*5pills） po. qd continue to disease progression plus XELOX (oxaliplatin 130mg/m2 d1; capecitabine 1000mg/m2 bid po. d1-14; q3w) or mFOLFOX (oxaliplatin 85mg/m2，d1; leucovorin 400mg/m2，d1；5-fluorouracil 400mg/m2，d1; 5-fluorouracil 2400mg/m2 continue 46h, q2w)
  Interventions: Drug: vitamin D3
- control group (Placebo Comparator): placebo 5 pills po. qd continue to disease progression plus XELOX (oxaliplatin 130mg/m2 d1; capecitabine 1000mg/m2 bid po. d1-14; q3w) or mFOLFOX (oxaliplatin 85mg/m2，d1; leucovorin 400mg/m2，d1；5-fluorouracil 400mg/m2，d1; 5-fluorouracil 2400mg/m2 continue 46h, q2w)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vitamin D3 — vitamin D3 400IU*5pills po. qd continue to disease progression
  Arms: Vitamin D3 group
Drug: Placebo — placebo 5 pills po. qd continue to disease progression
  Arms: control group

SUMMARY:
The study is a randomized,multicenter, double-blinded,phase III study. To explore the affection of vitamin D3 in combination with oxaliplatin plus fluoropyrimidine versus oxaliplatin plus fluoropyrimidine as first-line chemotherapy in previously untreated advanced or metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* males and females, ≥18 years of age
* All subjects must have inoperable, advanced or metastatic colorectal cancer and have confirmed histologically adenocarcinoma.
* Subject must be previously untreated with systemic treatment given as primary therapy for advanced or metastatic disease.
* Prior adjuvant or neoadjuvant chemotherapy and/or radiotherapy are permitted as long as the last administration of the last regimen occurred at least 12 months prior to randomization.
* ECOG performance status score of 0 or 1.
* Subjects must have at least one measurable lesion or evaluable disease by CT of MRI per RECIST1.1 criteria.
* Screening laboratory values must meet the following criteria in 7days before the first day of cycle 1:

  1. Hemoglobin ≥9.0g/dL;
  2. Neutrophils ≥1500/mm3;
  3. Platelet ≥100,000/mm3;
  4. Total Bilirubin ≤1.5*ULN
  5. AST ≤2.5*ULN (or ≤5.0*ULN if liver metastases are present), and ALT ≤2.5*ULN (or ≤5.0*ULN if liver metastases are present)
  6. Serum creatinine ≤1.5*ULN or calculated creatinine clearance >50mL/min
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days before randomization. All subjects of childbearing potential must agree to follow instructions for method of contraception for the duration of study treatment and 6 months after the last dose of study treatment.
* Life expectancy ≥3 months.

Exclusion Criteria:

* Concurrent diseases:

  1. Prior malignancy active cancer except for locally curable cancer that have been cured over 5years,or carcinoma in situ.
  2. Known brain metastasis
  3. Any serious or uncontrolled medical disorder or active infection.
  4. Known history of positive test for HIV or AIDS;
  5. Hepatitis B virus or hepatitis C virus is active;
* Within 4 weeks before randomization had operation, enlarged area radiotherapy(local radiotherapy within 2weeks) and other study drugs.
* Subjects with ≥ Grade 2 peripheral neuropathy.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
PFS(progression-free survival) | 5 years
  PFS is defined the time from the date of randomization to the date of disease progression or death due to any cause.

SECONDARY OUTCOMES:
OS(overall survival) | 5 years
  OS is defined the time between the date of randomization and the date of death.
DCR | up to 1 year
  disease control rate
ORR | up to 1 year
  overall response rate
Incidence of Treatment-Emergent Adverse Events | through study completion, an average of 1 year
  all the adverse events

IPD SHARING:
Plan to Share IPD: No